CLINICAL TRIAL: NCT00709813
Title: Including Patient Preferences in Symptom Management of Cancer Patients: A Randomized Clinical Trial
Brief Title: Study to Test a Computer-assisted Support System to Improve Patient-centered Care and Symptom Relief in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Cornelia M. Ruland, Professor, Rikshospitalet-Radiumhospitalet HF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCN 154739/320
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-03

CONDITIONS: Cancer; Lymphoma; Leukemia; Stem Cell Transplantation
Keywords: Symptom management; Cancer; Patient-centered care
MeSH Terms: conditions — Neoplasms; Lymphoma; Leukemia | interventions — Nurses; Inosine Triphosphatase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Behavioral: Tailored assessments provided to physicians and nurses (CHOICE, the Computer-assisted Interactive Tailored Patient Assessment Tool (ITPA))

INTERVENTIONS:
Behavioral: Tailored assessments provided to physicians and nurses (CHOICE, the Computer-assisted Interactive Tailored Patient Assessment Tool (ITPA)) — Both groups used CHOICE, the Computer-assisted Interactive Tailored Patient Assessment Tool (ITPA)for symptom assessments at in- and outpatient visits during and up-to nine months after treatment. In the intervention group physicians and nurses had assessment summaries available for care planning, displaying patients' symptoms, problems and concerns in rank-order of their needs for care. In the control group assessments were not available to care providers at any time.
  Arms: 2

SUMMARY:
Patient-provider shared decision making and the inclusion of patients' illness experiences and preferences in patient care are prioritized areas in health care. CHOICE is a computer-based support system for patient-centered symptom management of cancer patients developed for this purpose. In this randomized clinical trial at Rikshospitalet- Radiumhospitalet HF 145 adult stem-cell transplantation and newly diagnosed lymphoma and leukemia patients used CHOICE for assessments of their symptoms, problems and priorities for care at in-and outpatient visits during treatment and rehabilitation. In the experimental group this information was shared with physicians an nurses for subsequent care planning, but not in the control group.

This study tested effects of CHOICE on symptom- related patient care and outcomes of symptom relief, patients' needs for care over time and patient satisfaction;(2) analyzed how patients' symptoms, needs for care varied during illness/treatment stages; and (3) evaluated CHOICE' ease of use and user satisfaction. Controlling for gender, age, diagnosis, and type/stage of treatment, education, depression, health related quality of life, and social support, repeated measurement models were used to test differences and variations in outcome variables within and between groups and over time.

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* Starting treatment for a newly diagnosed acute myelogenous leukemia (AML), lymphatic leukemia (ALL), Hodgkin or non-Hodgkin lymphoma, or
* starting treatment for a recurrence of the disease;
* starting treatment with allogenous or autologous Stem Cell Transplantation (SCT).
* above 18 years of age.

Exclusion Criteria:

* having received radiation on the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Physicians' and nurses' symptom-related chart entries in patients' records | In-patient episodes of care
Symptom distress over time | Repeated episodes of care
Patients' prioritized needs for care over time | Repeated episodes of care

SECONDARY OUTCOMES:
Patient satisfaction | End of study
Care providers' satisfaction | End of study
Preferences for participation in decision making- and changes over time | Baseline, and at completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Rikshospitalet-Radiumhospitalet

REFERENCES:
- [Background] Ruland CM. Clinicians' perceived usefulness of a support system for patient-centered cancer care. Stud Health Technol Inform. 2006;124:624-30. PMID 17108586
- [Result] Ruland CM, Bakken S, Roislien J. Reliability and validity issues related to interactive tailored patient assessments: a case study. J Med Internet Res. 2007 Aug 1;9(3):e22. doi: 10.2196/jmir.9.3.e22. PMID 17942384